CLINICAL TRIAL: NCT03011073
Title: Evaluation of New Items in Cardiac Echography
Acronym: EPIC
Status: Withdrawn | Type: Observational
Why Stopped: investigator decision
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-09

CONDITIONS: Cardiac Echography; Cardiac Ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Paris Saint Joseph hospital has just acquired a new echocardiography EPIC . This new system has image processing and left ventricular function quantification software which are different from the precedent model Philips IE33.Left ventricular function quantification and myocardial distortion are the main medical examination influencing doctor's decisions.

EPIC can evaluate and quantify the cardiac ejection fraction via new software. Myocardial distortion quantification software also has been modified with new cut off and different calculation method.

The aim of this study is to compare the quality of images and the quantification of cardiac ejection fraction with these new software in order to choose the more reliable and reproducible for patient.

ELIGIBILITY:
Inclusion Criteria:

* patient accepting to stay 15 min more
* Age > 18 years old

Exclusion Criteria:

* patient not accepting this procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient who have prescription to do an cardiac ultrasound
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-10-06 (Estimated)

PRIMARY OUTCOMES:
Cardiac left ejection fraction | Day 1
  Evaluation of left ejection fraction by 3D

SECONDARY OUTCOMES:
Echographic images evaluation | day 1

IPD SHARING:
Plan to Share IPD: No